CLINICAL TRIAL: NCT00397631
Title: A Multicenter, Randomized, Double-Blind Study to Evaluate the Safety and Efficacy of the Initial Therapy With Coadministration of Sitagliptin and Pioglitazone in Patients With Type 2 Diabetes Mellitus
Brief Title: Initial Combination With Pioglitazone Study (0431-064)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-064; MK0431-064; 2006_531
Record Dates: First submitted 2006-11-08; First posted 2006-11-09 (Estimated); Results first posted 2009-07-10 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): sitagliptin 100 mg q.d./pioglitazone 30 mg q.d.
  Interventions: Drug: sitagliptin 100 mg q.d./pioglitazone 30 mg q.d
- 2 (Active Comparator): sitagliptin 100 mg placebo q.d./pioglitazone 30 mg q.d.
  Interventions: Drug: Comparator: placebo to match sitagliptin 100 mg q.d./pioglitazone 30 mg q.d.

INTERVENTIONS:
Drug: sitagliptin 100 mg q.d./pioglitazone 30 mg q.d — Patients will receive initial combination therapy with blinded sitagliptin 100 mg q.d. and open- label pioglitazone 30 mg q.d. for up to 24 Weeks. Sitagliptin 100 mg q.d. and pioglitazone 30 mg q.d. will be administered as oral tablets.
  Arms: 1
Drug: Comparator: placebo to match sitagliptin 100 mg q.d./pioglitazone 30 mg q.d. — Patients will receive placebo to match sitagliptin 100 mg q.d. (blinded) and open label pioglitazone 30 mg q.d. for up to 24 Weeks. Placebo to match sitagliptin 100 mg q.d.(blinded) and open-label pioglitazone 30 mg q.d. will be administered as oral tablets.
  Arms: 2

SUMMARY:
A clinical study to evaluate the safety and efficacy of the initial combination therapy with sitagliptin and pioglitazone in patients with type 2 diabetes mellitus not on treatment with insulin or oral antihyperglycemic therapy.

ELIGIBILITY:
General Inclusion Criteria:

* Patients ≥18 years old with Type 2 Diabetes Mellitus (a specific type of diabetes)

General Exclusion Criteria:

* Patient has a history of type 1 diabetes mellitus or history of ketoacidosis
* Patient was on antihyperglycemic agent therapy (oral or insulin) within the prior 4 months
* Patient was on >4 weeks (cumulatively) of antihyperglycemic therapy (oral or insulin) over the prior 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Actual)
Dates: Start 2006-12-19 (Actual); Primary Completion 2008-06-28 (Actual); Study Completion 2008-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Yoon KH, Shockey GR, Teng R, Golm GT, Thakkar PR, Meehan AG, Williams-Herman DE, Kaufman KD, Amatruda JM, Steinberg H. Effect of initial combination therapy with sitagliptin, a dipeptidyl peptidase-4 inhibitor, and pioglitazone on glycemic control and measures of beta-cell function in patients with type 2 diabetes. Int J Clin Pract. 2011 Feb;65(2):154-64. doi: 10.1111/j.1742-1241.2010.02589.x. PMID 21235696
- [Derived] Yoon KH, Steinberg H, Teng R, Golm GT, Lee M, O'Neill EA, Kaufman KD, Goldstein BJ. Efficacy and safety of initial combination therapy with sitagliptin and pioglitazone in patients with type 2 diabetes: a 54-week study. Diabetes Obes Metab. 2012 Aug;14(8):745-52. doi: 10.1111/j.1463-1326.2012.01594.x. Epub 2012 Apr 17. PMID 22405352

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Patient In: 01-Feb-2007; Last Patient Last Visit: 28-Jun-2008; 60 study sites worldwide.
Pre-assignment Details: Patients ≥18 years of age with type 2 diabetes mellitus (T2DM) with inadequate glycemic control (HbA1C
  ≥8% and ≤12%) on diet and exercise alone were eligible for randomization.
Groups:
- Sitagliptin 100 mg q.d. + Pioglitazone 30 mg q.d.: The Sitagliptin 100 mg q.d. + Pioglitazone 30 mg q.d. (q.d. = once daily) group includes data from patients randomized to receive coadministration of sitagliptin 100 mg oral tablets and pioglitazone 30 mg oral tablets administered once daily.
- Pioglitazone 30 mg q.d.: The Pioglitazone 30 mg q.d. (q.d. = once daily) group includes data from patients randomized to receive coadministration of pioglitazone 30 mg oral tablets and placebo to sitagliptin 100 mg oral tablets administered once daily.
Period: Overall Study
Arm/Group | Sitagliptin 100 mg q.d. + Pioglitazone 30 mg q.d. | Pioglitazone 30 mg q.d.
Started | 261 (Randomization ratio was 1:1) | 259
Completed | 231 | 215
Not Completed | 30 | 44
Not completed — Adverse Event | 5 | 6
Not completed — Lack of Efficacy | 7 | 10
Not completed — Lost to Follow-up | 8 | 9
Not completed — Physician Decision | 2 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 7 | 14
Not completed — protocol discontinuation criteria | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin 100 mg q.d. + Pioglitazone 30 mg q.d. | Pioglitazone 30 mg q.d. | Total
Number analyzed (Participants) | 261 | 259 | 520
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (10.2) | 51.6 (11.2) | 50.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 114 | 238
  Male | 137 | 145 | 282
Race/Ethnicity, Customized [Number; unit: participants]
  White | 138 | 134 | 272
  Black | 11 | 8 | 19
  Asian | 85 | 83 | 168
  Other | 27 | 34 | 61
HbA1c (Hemoglobin A1C) [Mean (Standard Deviation); unit: Percent] | 9.5 (1.2) | 9.5 (1.2) | 9.5 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (Hemoglobin A1C) at Week 24
Description: HbA1c is measured as a percent. Thus, this change from baseline reflects the Week 24 HbA1c percent minus the Week 0 HbA1c percent.
Time Frame: Baseline and 24 weeks
Population: The Full Analysis Set (FAS) included all patients with a baseline value and ≥1 post-baseline value for this outcome. For FAS patients with no data at Week 24, the last observed measurement was carried forward to Week 24.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Sitagliptin 100 mg q.d. + Pioglitazone 30 mg q.d. | Pioglitazone 30 mg q.d.
Number analyzed (Participants) | 251 | 246
Percent | -2.38 [-2.55 to -2.21] | -1.49 [-1.66 to -1.32]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg q.d. + Pioglitazone 30 mg q.d. vs Pioglitazone 30 mg q.d; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, baseline HbA1c; Mean Difference (Net) = -0.89, 95% CI [-1.13 to -0.65], Standard Error of Mean 0.12

2. Secondary Outcome: Change From Baseline in FPG (Fasting Plasma Glucose) at Week 24
Description: Change from baseline at Week 24 is defined as Week 24 minus Week 0.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg q.d. + Pioglitazone 30 mg q.d. | Pioglitazone 30 mg q.d.
Number analyzed (Participants) | 256 | 253
mg/dL | -63.0 [-68.3 to -57.6] | -40.2 [-45.6 to -34.8]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg q.d. + Pioglitazone 30 mg q.d. vs Pioglitazone 30 mg q.d; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, baseline FPG; Mean Difference (Net) = -22.8, 95% CI [-30.4 to -15.2], Standard Error of Mean 3.87

3. Secondary Outcome: Change From Baseline in 2-hour PPG (Post-prandial Glucose) at Week 24
Description: Change from baseline at Week 24 is defined as Week 24 minus Week 0.
Time Frame: Baseline and Week 24
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin 100 mg q.d. + Pioglitazone 30 mg q.d. | Pioglitazone 30 mg q.d.
Number analyzed (Participants) | 216 | 211
mg/dL | -113.6 [-122.4 to -104.8] | -68.9 [-77.8 to -60.0]
Statistical Analysis 1: Comparison: Sitagliptin 100 mg q.d. + Pioglitazone 30 mg q.d. vs Pioglitazone 30 mg q.d; Test type: Superiority or Other; p < 0.001, ANCOVA; Model terms: treatment, baseline 2-hour PPG; Mean Difference (Net) = -44.7, 95% CI [-57.2 to 32.2], Standard Error of Mean 6.37

ADVERSE EVENTS:
Arm/Group | Sitagliptin 100 mg q.d. + Pioglitazone 30 mg q.d. | Pioglitazone 30 mg q.d.
Serious Adverse Events (participants affected / at risk) | 8 | 5
Other Adverse Events (participants affected / at risk) | 17 | 25
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Sitagliptin 100 mg q.d. + Pioglitazone 30 mg q.d. | Pioglitazone 30 mg q.d.
Any Ear and labyrinth disorders (Ear and labyrinth disorders) | 1/261 | 0/259
Acute vestibular syndrome (Ear and labyrinth disorders) | 1/261 | 0/259
Any Gastrointestinal disorders (Gastrointestinal disorders) | 2/261 | 0/259
Abdominal pain upper (Gastrointestinal disorders) | 1/261 | 0/259
Peptic ulcer (Gastrointestinal disorders) | 1/261 | 0/259
Any Infections and infestations (Infections and infestations) | 2/261 | 1/259
Abscess limb (Infections and infestations) | 0/261 | 1/259
Bronchitis bacterial (Infections and infestations) | 1/261 | 0/259
Pulmonary tuberculosis (Infections and infestations) | 1/261 | 0/259
Any Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 1/261 | 1/259
Foreign body trauma (Injury, poisoning and procedural complications) | 0/261 | 1/259
Humerus fracture (Injury, poisoning and procedural complications) | 1/261 | 0/259
Any Nervous system disorders (Nervous system disorders) | 0/261 | 2/259
Cerebrovascular accident (Nervous system disorders) | 0/261 | 1/259
Transient ischaemic attack (Nervous system disorders) | 0/261 | 1/259
Any Psychiatric disorders (Psychiatric disorders) | 1/261 | 0/259
Impulsive behaviour (Psychiatric disorders) | 1/261 | 0/259
Any Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 1/261 | 0/259
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 1/261 | 0/259
Any Vascular disorders (Vascular disorders) | 0/261 | 1/259
Peripheral ischaemia (Vascular disorders) | 0/261 | 1/259
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Sitagliptin 100 mg q.d. + Pioglitazone 30 mg q.d. | Pioglitazone 30 mg q.d.
Any Infections and infestations (Infections and infestations) | 8/261 | 14/259
Nasopharyngitis (Infections and infestations) | 8/261 | 14/259
Any Nervous system disorders (Nervous system disorders) | 9/261 | 13/259
Headache (Nervous system disorders) | 9/261 | 13/259

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.